CLINICAL TRIAL: NCT00473447
Title: Phase1 Effectiveness of a Modified Constraint-Induced Movement Therapy Program in Rehabilitation of Arm Paresis in Children With Cerebral Palsy: a Cross-Over Study
Brief Title: A Modified Constraint-Induced Movement Therapy Program in Rehabilitation of Arm Paresis in Children With Cerebral Palsy
Acronym: mCIT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universita di Verona (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 800
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Last update posted 2007-05-15 (Estimated); Status verified 2007-05

CONDITIONS: Hemiparesis; Cerebral Palsy
Keywords: Rehabilitation; Children; Cerebral Palsy; Arm; Paresis
MeSH Terms: conditions — Paresis; Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Modified Constraint-induced movement therapy

SUMMARY:
The purpose of this study is to determine if a modified protocol of constraint-induced movement therapy (CIT) is effective in rehabilitation treatment of arm paresis in children with cerebral palsy. In these children one main problem the non-use of the affected arm. Many studies showed that the non-use phenomenon can by reversed by the CIT, a rehabilitation program consisting of 15 days of restraining the unaffected arm plus a daily intensive (6 hours/day) physiotherapy training of the paretic arm. The present study aims at evaluating if a shortened CIT protocol (restraining device plus only 2 weekly hours of physiotherapy) is effective in improving use and function of children paretic arm

ELIGIBILITY:
Inclusion Criteria:

* presence of mild-moderate arm paresis (after cerebral palsy) enabling to
* reach and grasp a pellet
* age between 1-10 years
* active participation during proposed activities
* parents consent for participation -

Exclusion Criteria:

* presence of severe behaviour disturbances
* presence of severe mental retardation (QI<60)

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2004-01; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Arm Use Test | Four months for each patient

SECONDARY OUTCOMES:
Arm Function Test | Four months for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Fiaschi, MD PhD, Study Director — Department of Neurological and Vision Sciences, University of Verona